CLINICAL TRIAL: NCT05957731
Title: Effect of Agonist Contract Relax Versus Antagonist Contract Relax Technique on Spasticity and Ankle Range of Motion in Chronic Stroke Patient.
Brief Title: Effect of Agonist Contract Relax Versus Antagonist Contract Relax in Chronic Stroke Patient.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-246-04-2023
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: Stroke; Agonist contract relax; antagonist contract relax; stretching; modified A
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Agonist Contract-relax group: (Experimental): In the agonist contract-relax group, participants were positioned in a supine position. A trained physiotherapist then passively dorsiflexed the ankle to its maximum available range and held it for 15 seconds, while ensuring that the knee remained straight by placing a hand on it. Following this, participants were instructed to perform a maximal voluntary isometric
  35
  contraction of the planter flexors for five seconds, while maintaining the stretched position.
  After a 30-second rest period, the physiotherapist returned the ankle to the starting position of 0 degrees and repeat the procedure without any rest. This stretching protocol was repeated four times, with each repetition lasting 2 minutes. For the soleus muscles, the same procedure was performed, but with a slightly flexed initial position of the knee.
  Interventions: Other: Routine physical therapy; Other: agonist contract relax
- Antagonist contract-relax group: (Experimental): In the antagonist stretching groups, participants were positioned in a supine position. A trained physiotherapist stretched the antagonist's muscle, and then participants were instructed to perform a maximal voluntary isometric contraction of dorsiflexion for 5 seconds while maintaining a stretched position. The knee was kept straight during this contraction.
  Following the contraction, the physiotherapist held the ankle at that angle for another 10 seconds by placing a hand on it. After a 30-second rest period, the physiotherapist returned the ankle to the starting position of 0 degrees and repeat the procedure without any rest intervals.
  Interventions: Other: Routine physical therapy; Other: antagonist contract relax

INTERVENTIONS:
Other: Routine physical therapy — Both groups received routine physical therapy, which encompasses various components such as electrotherapy, strength training for both lower and upper limbs, gait training, and occupational therapy.
Other: antagonist contract relax — antagonist contraction i used to improve spasticity and range of motion in stroke patients
  Arms: Antagonist contract-relax group:
Other: agonist contract relax — agonist contraction is used to improve spasticity and range of motion in stroke patients
  Other Names: agonist contraction
  Arms: Agonist Contract-relax group:

SUMMARY:
It will be a randomized control trial with 112 patients which will be divided into two groups of 56 patients in each group. Participants will recruit through convenient sampling techniques.

Outcome measures are range of motion and spasticity. The protocol was implemented three days per week for eight consecutive weeks. Data will be collected at baseline and 8 th week after intervention.

DETAILED DESCRIPTION:
Objective of the study is to compare the effects of the agonist contract-relax technique versus the antagonist contract-relax technique on spasticity and range of motion in individuals with chronic stroke.

Null hypothesis (H0):

There are no comparative effects of agonist contact-relax technique and the antagonist contract-relax technique on spasticity and ankle range of motion in chronic patients.

The alternate hypothesis (HA):

There are comparative effects of agonist contract-relax technique and the antagonist contract-relax technique on spasticity and ankle range of motion in chronic stroke patients.

The sample size came out to 94 (47 in each group) after adding 20% dropout the sample size was 47+9=56 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of stroke by a neurologist.
* Inclusion of patients with both ischemic and hemorrhagic stroke.
* Both male and female patients are eligible.
* Age range between 40 to 60 years.
* Modified Ashworth Scale ranging from 0 to 2.
* Minimum muscle strength grade of 3

Exclusion Criteria:

* History of surgery on lower limb
* Who received injection therapies for reducing spasticity
* Lower extremity contracture
* Modified Ashworth scale of 3-4

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale. | it will measure change in spasticity at baseline and at 8th week
  The assessment involves extending the limb of the parent from a state of utmost flexion to utmost extension, identifying the point at which initial mild resistance was encountered. Following that, the modified Ashworth Scale is employed while transitioning the limb from extension to flexion. Interrater reliability studies utilizing the MAS have yielded varied results, ranging from moderate to good.
universal goniometer | it will measure change in range of motion at baseline and at 8th week
  The universal goniometer (UG) is a widely employed tool for assessing range of motion.Range of motion refers to the complete extent of movement possible at a specific joint. In a normal ankle, the range of motion typically spans from around 20ºof dorsiflexion to 50º of plantar flexion. For normal walking, a combined motion of approximately 24º to 30º (including both dorsiflexion and plantar flexion) is required.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - sir Ganga Raam hospital lahore, Lahore
  - univerity of Lahore teaching hopital, Lahore

IPD SHARING:
Plan to Share IPD: No